CLINICAL TRIAL: NCT04830163
Title: Upregulating Corticospinal Function After Stroke Using Brain State-dependent Paired Corticomotoneuronal Stimulation
Brief Title: Brain State-dependent PCMS in Chronic Stroke
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000896_Exp3
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: chronic, movement
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCMS during brain states reflecting strong corticospinal transmission (Experimental)
  Interventions: Combination Product: Brain state-dependent paired corticomotoneuronal stimulation (PCMS)
- PCMS during random brain states (Active Comparator)
  Interventions: Combination Product: Brain state-dependent paired corticomotoneuronal stimulation (PCMS)

INTERVENTIONS:
Combination Product: Brain state-dependent paired corticomotoneuronal stimulation (PCMS) — Paired corticomotoneuronal stimulation (PCMS) involves delivering precisely timed pairs of transcranial magnetic stimulation (TMS) and peripheral nerve stimulation (PNS) so that the neuronal activity evoked by such stimulation arrives synchronously at corticospinal-motoneuronal synapses. This synchronous arrival is postulated to cause long-term potentiation via spike timing-dependent plasticity, which then improves corticospinal transmission and hand function. In this study, paired corticomotoneuronal stimulation (PCMS) will be applied during specific brain states that reflect increased recruitment of motoneurons via the corticospinal tract. This increased recruitment is expected to enhance the beneficial effects of PCMS on human hand function after stroke.

SUMMARY:
After stroke, people often have difficulty using their hands. Combined brain and nerve stimulation can strengthen the neural pathways that control hand function. In this study, we will deliver combined brain and nerve stimulation during specific time windows that increase activation of neural pathways underlying hand function. We will compare the effects of combined brain and nerve stimulation during these optimal time windows to the effects of combined brain and nerve stimulation applied during random time windows on post-stroke hand function.

ELIGIBILITY:
Inclusion Criteria:

* History of stroke > 6 months ago
* Presence of residual upper extremity hemiparesis
* Willingness to participate
* Ability to provide informed consent
* Upper extremity Fugl-Meyer score < 66
* Mini Mental State Exam score > 24
* Discernible and reliable motor-evoked potential (MEP) elicited following single-pulse TMS to the lesioned hemisphere

Exclusion Criteria:

* History of neurological disease other than stroke
* Presence of contraindications to transcranial magnetic stimulation (TMS) or peripheral nerve stimulation (PNS), including: history of adverse reactions to TMS or PNS metal in head, eyes, neck, chest/trunk, or arms, including but not limited to shrapnel, surgical clips, fragments from metalworking, fragments from welding, implanted device, history of frequent and severe headaches or migraines, immediate family history of seizure or epilepsy, personal history of seizure or epilepsy, current, suspected, or planned pregnancy, current or recent (within the last 3 months) use of medications acting on the central nervous system other than selective serotonin reuptake inhibitors (SSRIs), including but not limited to antipsychotic drugs, benzodiazepines, prescription stimulants.
* Upper extremity Fugl-Meyer score ≥ 66 (66 is the maximum on this scale)
* Mini Mental State Exam score <= 24
* No discernible and reliable MEP elicited following single-pulse TMS to the lesioned hemisphere

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Maximum hand force output | up to 1 hour after intervention
  This will be measured using maximum voluntary contractions of the stroke-affected first dorsal interosseous hand muscle during pinching actions.
Maximum hand muscle activation | up to 1 hour after intervention
  This will be measured using electromyography recordings of the stroke-affected first dorsal interosseous muscle during maximum voluntary contractions during pinching actions

SECONDARY OUTCOMES:
Amplitude of motor evoked potentials | up to 1 hour after intervention
  This will be measured as the peak-to-peak amplitude of motor-evoked potentials recorded from the stroke-affected first dorsal interosseous muscle
Time to complete the 9-hole peg test | up to 1 hour after intervention
  This will be measured as the time needed to complete the task using the stroke-affected hand.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be shared using an open-access data repository. No personally-identifiable information will be shared.